CLINICAL TRIAL: NCT04247412
Title: Laryngomicrosurgery Under Nonintubated Deep Paralysis (NIDP) General Anesthesia Supported by Transnasal Humidified Rapid-insufflation Ventilatory Exchange: A Case Series Study
Brief Title: Laryngomicrosurgery Under NIDP General Anesthesia Supported by THRIVE
Acronym: NIDP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Principal Investigator, RenJi Hospital
Other Study IDs: diansansu
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Vocal Polyp
Keywords: Laryngomicrosurgery; Nonintubated deep paralysis; Transnasal Humidified Rapid-insufflation Ventilatory Exchange

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laryngomicrosurgery requires deep paralysis and general anesthesia to finish the procedure. After the procedure, patients need a long time to recover. In the present study, with the support of the transnasal humidified rapid-insufflation ventilatory exchange, laryngomicrosurgery would be finished under nonintubated deep paralysis (NIDP) general anesthesia. In this case series study, the investigators will test the safety and feasibility of such a technique.

ELIGIBILITY:
Inclusion Criteria:

* elective polypectomy of unilateral vocal cord
* age between 18 to 40
* be able to communicate
* estimated operation time less than 15min
* ASA I-II
* Agree to sign written informed consent

Exclusion Criteria:

* pregnancy or breastfeeding women
* severe gastrointestinal reflex disease
* neuromuscular disease
* body mass index(BMI)>30
* predictable difficult airway.
* allergy to medicine would be used in the present study including propofol, remifentanil or sugammadex

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young patients who will under elective polypectomy of unilateral vocal cord.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of laryngomicrosurgery | From the day before surgery till 2 days after surgery or before discharge
  complete the surgery within 15min,nonintubated,remove the polyp entirely,recover completely after surgery, no major adverse event

SECONDARY OUTCOMES:
Total days that participants stay in hospital | Through study completion, an average 2 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fan Y, Chi X, Zhu D, Yin J, Liu Y, Su D. Non-intubated deep paralysis: a new anaesthesia strategy for vocal cord polypectomy. Perioper Med (Lond). 2023 Apr 19;12(1):12. doi: 10.1186/s13741-023-00301-7. PMID 37076883